CLINICAL TRIAL: NCT02163590
Title: A Preliminary Investigation Into the Immediate Effects of Different Rates of Thoracic Mobilization on Pressure Pain Thresholds in Asymptomatic Individuals
Brief Title: Immediate Effects of Different Rates of Thoracic Mobilization on Pressure Pain Thresholds in Asymptomatic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Francisco Xavier de Araujo, Pt, Physical therapist - Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFCSPA-FXA-02
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Spine Stiffness
Keywords: Spinal mobilisation; Pressure pain threshold; Thoracic spine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2Hz mobilisation (Experimental): A bilateral postero-anterior mobilisation applied to the fourth thoracic vertebra, at a 2Hz frequency.
  Interventions: Other: 2Hz mobilisation
- 0,5Hz mobilisation (Experimental): A bilateral postero-anterior mobilisation applied to the fourth thoracic vertebra, at a 0,5Hz frequency.
  Interventions: Other: 0,5Hz mobilisation
- Placebo (Placebo Comparator): A simulation technique, that mimic the other groups, in this case only manual contact will be applied, without any oscillation.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 2Hz mobilisation — This intervention will be applied for 3 sets of 1 minute, with 1 minute rest period in between each set.
  Other Names: Bilateral postero-anterior thoracic mobilisation
  Arms: 2Hz mobilisation
Other: 0,5Hz mobilisation — This intervention will be applied for 3 sets of 1 minute, with 1 minute rest period in between each set.
  Other Names: Bilateral postero-anterior thoracic mobilisation
  Arms: 0,5Hz mobilisation
Other: Placebo — Intervention that mimics the experimental procedures
  Other Names: Manual contact without oscillation
  Arms: Placebo

SUMMARY:
Passive mobilizations of the spine are widely used by physiotherapists in the management of neuromusculoskeletal disorders.

There is a nascent body of work of the mechanical properties of joint mobilizations. Treatment dose is characterized by the direction of force applied, magnitude of force applied, frequency of oscillation, amplitude of displacement, repetition and time. Although the choice of better treatment dose is based on patient complaints and clinical reasoning, the comprehension of the effects of different parameters of joint mobilization will improve the decision making process. The optimal dose of treatment, however, is not already known.

The primary aim of this study is to determine whether different rates of thoracic mobilization are capable to produces hypoalgesic effects, and secondarily investigate if such effects are local or widespread.

DETAILED DESCRIPTION:
Healthy volunteers will be recruited and randomized into 3 groups. A 2Hz mobilisation group, a 0,5Hz mobilisation group and a Placebo group. The pressure pain threshold will be measured before, immediately after and 15 minutes after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy asymptomatic subjects
* Manual therapy naive

Exclusion Criteria:

* Any kind of history of trauma or surgery to the spine
* Contraindications or precautions to manual therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Change from baseline imediately after, and 15 minutes after the intervention
  Pressure pain threshold will be measured in five anatomic points on the spine, upper and lower limbs

CONTACTS AND LOCATIONS:
Overall Officials: Francisco D Araujo, Pt, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil